CLINICAL TRIAL: NCT00016627
Title: Linkage Study in Familial Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 969; U01HL067467 (NIH)
Record Dates: First submitted 2001-05-19; First posted 2001-05-21 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-11

CONDITIONS: Pulmonary Fibrosis; Lung Diseases; Lung Diseases, Interstitial
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases; Lung Diseases, Interstitial

SUMMARY:
To map the gene (or genes) for familial pulmonary fibrosis.

DETAILED DESCRIPTION:
BACKGROUND:

Familial pulmonary fibrosis (FPF) is a rare, progressive, life-threatening disease. Although far from definitive, several lines of evidence suggest that it could involve genetic susceptibility and that its expression may be modified gene-environment interactions involving exposure to fibrogenic dusts. If the specific gene loci involved can be identified and their functions characterized, these studies could lead to a better understanding of the etiology of the disease and effective intervention strategies among families at increased risk. It is conceivable that the genetically influenced pathologic mechanisms involved may be shared with other, more common forms of pulmonary fibrosis such as idiopathic pulmonary fibrosis (IPF) or asbestosis. Thus, these studies could lead to the early identification of individuals susceptible to reversible interstitial lung disease and to the development of novel therapeutic approaches.

Familial pulmonary fibrosis is indistinguishable pathologically from idiopathic pulmonary fibrosis and appears to be inherited as an autosomal dominant trait with variable penetrance; pulmonary fibrosis is associated with pleiotropic genetic disorders, such as Hermansky-Pudlak syndrome, neurofibromatosis, tuberous sclerosis, Neimann-Pick disease, Gaucher's disease, and familial hypocalciuric hypercalcemia; pulmonary fibrosis is frequently observed in autoimmune disease, including rheumatoid arthritis and systemic sclerosis; variable susceptibility is evident among workers who are reported to be exposed occupationally to similar concentrations of fibrogenic dusts; and inbred strains of mice differ in their susceptibility to fibrogenic dust.

DESIGN NARRATIVE:

The study uses standard genetic methodology (linkage analysis) to investigate the distribution of polymorphisms for anonymous genetic markers in families with familial pulmonary fibrosis. The comprehensive genome-wide study, using standard genetic markers, will allow identification of loci which subsequently may prove to contain novel genes that play a role in the pathogenesis of pulmonary fibrosis. Once genetic loci are defined in familial pulmonary fibrosis, candidate genes can be identified on the basis of both positional and functional criteria. Moreover, this approach will provide basic information on high priority loci that will be applicable to the rapidly evolving dense human transcript map for pulmonary fibrosis in families with two or more cases of pulmonary fibrosis.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Steele — Duke University

REFERENCES:
- [Background] Wahidi MM, Speer MC, Steele MP, Brown KK, Schwarz MI, Schwartz DA. Familial pulmonary fibrosis in the United States. Chest. 2002 Mar;121(3 Suppl):30S. doi: 10.1378/chest.121.3_suppl.30s. No abstract available. PMID 11893669
- [Background] Savov JD, Brass DM, Berman KG, McElvania E, Schwartz DA. Fibrinolysis in LPS-induced chronic airway disease. Am J Physiol Lung Cell Mol Physiol. 2003 Oct;285(4):L940-8. doi: 10.1152/ajplung.00102.2003. Epub 2003 Jun 20. PMID 12818888
- [Background] Garantziotis S, Steele MP, Schwartz DA. Pulmonary fibrosis: thinking outside of the lung. J Clin Invest. 2004 Aug;114(3):319-21. doi: 10.1172/JCI22497. PMID 15286797
- [Background] Steele MP, Speer MC, Loyd JE, Brown KK, Herron A, Slifer SH, Burch LH, Wahidi MM, Phillips JA 3rd, Sporn TA, McAdams HP, Schwarz MI, Schwartz DA. Clinical and pathologic features of familial interstitial pneumonia. Am J Respir Crit Care Med. 2005 Nov 1;172(9):1146-52. doi: 10.1164/rccm.200408-1104OC. Epub 2005 Aug 18. PMID 16109978
- [Derived] Garantziotis S, Zudaire E, Trempus CS, Hollingsworth JW, Jiang D, Lancaster LH, Richardson E, Zhuo L, Cuttitta F, Brown KK, Noble PW, Kimata K, Schwartz DA. Serum inter-alpha-trypsin inhibitor and matrix hyaluronan promote angiogenesis in fibrotic lung injury. Am J Respir Crit Care Med. 2008 Nov 1;178(9):939-47. doi: 10.1164/rccm.200803-386OC. Epub 2008 Aug 14. PMID 18703791